CLINICAL TRIAL: NCT07254104
Title: Clinical Evaluation of [68Ga]Ga-NOTA-RF PET Imaging Targeting RFVT3 in Patients With Pituitary Tumors
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xianzhong Zhang, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-RFVT3
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pituitary Neoplasms
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pituitary Neoplasms (Experimental): Participants with pituitary neoplasms will undergo [68Ga]Ga-NOTA-RF PET/CT imaging to evaluate tracer uptake, biodistribution, and safety.
  Interventions: Drug: [68Ga]Ga-NOTA-RF

INTERVENTIONS:
Drug: [68Ga]Ga-NOTA-RF — Administer the [68Ga]Ga-NOTA-RF radiotracer via injection.
  Other Names: [68Ga]Ga-RF PET tracer

SUMMARY:
This study aims to evaluate the clinical application value of [68Ga]Ga-NOTA-RF, a novel PET molecular probe targeting riboflavin transporter 3 (RFVT3), in patients with pituitary adenomas. It will observe the probe's imaging characteristics, distribution signs, and the relationships between these factors, tumor differentiation degree, and radiotracer uptake. Additionally, the study will explore the diagnostic advantages of [68Ga]Ga-NOTA-RF in patients with pituitary adenomas and its potential value in precise typing.

DETAILED DESCRIPTION:
This study aims to evaluate the potential clinical application of [68Ga]Ga-NOTA-RF in pituitary adenomas. Such tumors are characterized by variable degrees of differentiation, subtle early morphological changes, complex metabolic states, and a strong dependence on mitochondrial activity. Existing imaging modalities have limited performance in detecting and characterizing these lesions, highlighting the need for novel metabolic imaging tools. This study will systematically investigate the biodistribution and imaging characteristics of [68Ga]Ga-NOTA-RF in pituitary adenomas, as well as its correlation with RFVT3 expression, to explore its potential value in early tumor detection, metabolic subtype differentiation, and molecular classification.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, male or female.
2. Able to understand and sign written informed consent, willing to follow pre-injection preparation requirements (adequate hydration and avoidance of high-dose riboflavin supplements), and to complete all study procedures.
3. Recurrent invasive pituitary adenoma within 6 months after surgery, without intracranial or distant metastasis. The postoperative pathological Ki-67 index of the previous pituitary tumor is ≥3%, and tumor growth cannot be controlled by standard medical therapy and radiotherapy.
4. Radiological and clinical evidence indicates residual or recurrent pituitary adenoma requiring treatment or follow-up management.
5. At least one measurable and resectable lesion suitable for correlation with PET imaging evaluation; vital signs are stable, and the participant is able to lie supine and cooperate during a 30-60 minute PET scan.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, or breastfeeding women.
2. Known history of severe allergic or anaphylactoid reactions to any component of the investigational tracer (riboflavin derivatives, NOTA chelator, or formulation excipients).
3. Presence of severe or uncontrolled medical conditions (e.g., decompensated heart failure, active infection, myocardial infarction or stroke within the past 4 weeks) that, in the opinion of the investigator, make the participant unsuitable for PET imaging.
4. Concomitant severe systemic diseases such as cardiac, pulmonary, hepatic, or renal failure.
5. Pituitary adenoma patients who underwent surgery less than 4 weeks prior to enrollment or completed radiotherapy to the sellar region within the past 3 months.
6. Participation in another interventional clinical trial within the past 4 weeks, or cumulative radiation exposure from prior research procedures within the past 12 months that may exceed the ethical safety limit.
7. Severe claustrophobia unrelieved by sedation, or any other condition that would prevent completion of the PET scan.
8. Poor compliance or any factor judged by the investigator to affect the participant's safety or the quality of study data.
9. Any other condition that, in the judgment of the investigator, makes the participant unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
SUVmax | After the completion of the PET examination.
  The tumor uptake capacity (expressed as SUV values) of [68Ga]Ga-NOTA-RF PET imaging in intracranial tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Xianzhong Zhang, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No